CLINICAL TRIAL: NCT07003906
Title: Treating Emergency Laparotomy Incisions With Negative Pressure Wound Therapy
Acronym: TELIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala County Council, Sweden (Other Government); Dalarna County Council, Sweden (Other); Sormland County Council, Sweden (Other); Ostergotland County Council, Sweden (Other); Västmanland County Council, Sweden (Other Government); Landstingens Ömsesidiga Försäkringsbolag (Löf) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TELIN-1337; CIV-24-11-049998 (Other: Swedish Medical Products Agency); FOU2025-00096 (Other: Uppsala County)
Record Dates: First submitted 2025-05-14; First posted 2025-06-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Surgical Incision; Wound Dehiscence; Surgical Site Infection; Incisional Hernia; Quality of Life
Keywords: emergency surgery; negative pressure wound therapy; randomised controlled trial
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection; Incisional Hernia | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments and analyses will be masked. It's not feasible to blind Participants and Care Providers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational device (Experimental): Will recieve 7 days of treatment with negative pressure wound therapy after closure of emergency surgery incision
  Interventions: Device: Negative pressure wound therapy
- Standard of care (Active Comparator): Will recieve a regular dressing after closure of emergency surgery incision
  Interventions: Device: Standard postoperative dressing

INTERVENTIONS:
Device: Negative pressure wound therapy — Avance Solo Negative Pressure Wound Therapy (NPWT) System is a portable battery powered single use negative pressure system, suitable for use in closed incision and chronic wound indications.
  The system consists of Avance Solo Pump, Avance Solo Canister 50 mL, Avance Solo Border Dressing and Avance Solo Foam.
  Other Names: Avance Solo
  Arms: Investigational device
Device: Standard postoperative dressing — Mepilex Border Post-Op is a self-adhesive absorbent surgical dressing designed for exuding wounds. It is intended for acute wounds, such as surgical wounds, cuts and abrasions.
  Other Names: Mepilex Border Post-Op
  Arms: Standard of care

SUMMARY:
The goal of this clinical trial is to investigate Negative Pressure Wound Therapy (NPWT) in adults undergoing emergency laparotomy. The main question it aims to answer is:

Does NPWT decrease wound complications?

Researchers will compare it against regular dressings to see if NPWT is superior.

DETAILED DESCRIPTION:
Negative Pressure Wound Therapy (NPWT) is a method of treating wounds using suction. The dressing is airtight, and the pump creates subatmospheric pressure, clearing the wound of exudate and fluids.

The study aims to investigate the effect of Negative pressure wound therapy dressings on the rate of wound complications (SSI, WD, seroma) after emergency laparotomy. Patients will be randomised to regular dressings and investigational device 1:1. No other aspect of the care will be changed.

Randomisation is planned at the time of skin closure. Patients will be followed-up after 7, 30 and 365 days with two initial visits, surveys and offered a CT scan to investigate incisional hernia formation.

The hypothesis is that NPWT dressings decrease the rate of wound complications. The secondary outcome is reduction of SSI, WD, seroma, shorter length of stay, peri-wound blistering, patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Written informed consent
* >10 cm midline incision with primary skin closure
* Emergency laparotomy

Exclusion Criteria:

* Not able to consent (e.g. dementia, impaired cognitive function, unconscious)
* Subjects not possible to follow up as assessed by the Investigator
* Allergy to dressing material
* Pregnancy or breastfeeding (females of childbearing potential)
* Previous enrolment in the current study
* Expected reoperation with 28 days of index laparotomy
* Emergency laparotomy within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Wound complications | 7 and 30 days
  Incident rate of wound complications (infection, dehiscence, seroma)

SECONDARY OUTCOMES:
Surgical site infections | 7 and 30 days
Wound dehiscence | 7 and 30 days
  Rupture of skin or fascia assessed clinically or with radiology.
Length of stay | 30 days
Quality of life survey | 30 days and 1 year
  EuroQoL Scale with 5 dimensions and 5 levels (EQ5D-5L). Patients scores in each dimension and total score indexed score is calculated where higher is better quality of life. Scores are weighted using published population values where 1 equals full health and worse health states goes towards, but can not reach 0. The EQ5D-5L also includes a VAS scale 0-100 where 100 is the best imaginable health and 0 the worst.
Scar satisfaction | 30 days and 1 year
  Patient and Observer Scar Assessment Scale (POSAS 2.0). Includes pain, vascularity, pigmentation, thickness, relief, pliability and surface area. Lower total score is better. The scale goes from 6-60 for patients and 6-60 for observers. Both also estimate an overall score 1-10 which is not included in the total score when using that aspect of the POSAS.
Incidence of incisional hernias | 1 year
  The incidence rate of incisional hernia, the measure is assessed by computer tomography, the need for surgery and clinical diagnosis
Mortality | 7, 30 days and 1 year
Costs | 30 days
  Cost of dressing and health care
Incidence of hernias | 5 years
  Hernia surgery and diagnoses from the National Patient Registry.
Incidence of small bowel obstruction | 5 years
  Small bowel obstruction surgery and diagnoses from the National Patient Registry.
Incidence of reconstructive surgery | 5 years
  Reconstructive abdominal wall surgery from the National Patient Registry.
Incidence rate of seromas | 7 and 30 days
  Seroma, i.e. collection of fluid in the subcutaneous tissue.
Incidence of hematomas | 7 and 30 days
  Hematoma, a collection of blood in the subcutaneous tissues.
Incidence of ischemia around and in wound | 7 and 30 days
  Composite measure of ischemia, necrosisis in wound
Incidence of enterocutaneus fistula | 7 and 30 days
  Enterocutaneous fistula formation
Need for antibiotics after surgery | 7 and 30 days
  Incidence rate of antibiotic treatment
Incidence of other infections after surgery | 7 and 30 days
  Composite measure of other infections (e.g., deep abdominal infections, urinary tract infections, pneumonia)
Number of healthcare visits after surgery | 7 and 30 days
  Number of healthcare visits
Reoperation rate | 7 and 30 days
  Any unscheduled surgery after first surgery

CONTACTS AND LOCATIONS:
Locations (6):
- Sweden (6):
  - Mälar Hospital, Eskilstuna
  - Linköping University Hospital, Linköping
  - Mora Hospital, Mora
  - Vrinnevi Hospital, Norrköping
  - Uppsala University Hospital, Uppsala
  - Västmanlands Hospital Västerås, Västerås

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data with complete removal of identifying information is planned to be available on request.